CLINICAL TRIAL: NCT01599455
Title: Cardiovascular Measurements at Baseline and During Cystometry in Pediatric Spinal Cord Injury
Brief Title: Baseline Cardiovascular Measurements in Pediatric Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Kathy Zebracki, Clinical Psychologist, Director of Psychology, Shriners Hospitals for Children
Other Study IDs: SHC-SCI-CV
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injury
Keywords: pediatric spinal cord injury; blood pressure; heart rate; baseline
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Inpatient: Youths admitted for inpatient rehabilitation training
- Outpatient: Youths visiting outpatient clinics
- Urodynamic study: Youths who undergo scheduled urodynamic study

SUMMARY:
Following spinal cord injury (SCI), the body loses normal control of blood pressure and heart rate, and there is a risk of sudden and dangerous increases in blood pressure, namely, autonomic dysreflexia (AD). It is important to be aware of baseline blood pressures and heart rates in individuals in order to detect AD. However, baseline values vary in developing children, and may be more variable in children with SCI. Thus, the objective of this study is to determine baseline blood pressure and heart rate measurements in children with SCI during rest and during urodynamic testing.

The investigators hypothesize that 1) blood pressures will increase with increasing age and body mass index; 2) heart rate will decrease with increasing age; 3) blood pressures will increase with increase in bladder filling; 4) blood pressures will increase will increase with increasing duration of injury.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents with spinal cord injury
* age 18 years or younger

Exclusion Criteria:

* known history of hypertension, cardiac, renal, or thyroid disease
* recent surgical procedure less than 2 weeks prior to admission or visit
* fever or signs of active infection or inflammation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with spinal cord injury who are admitted for spinal cord injury rehabilitation program, visiting outpatient clinics, or undergoing scheduled urodynamic study
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2012-05; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure readings | at regularly scheduled medical appointments

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospitals for Children - Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zebracki K, Hwang M, Patt PL, Vogel LC. Autonomic cardiovascular dysfunction and vitamin D deficiency in pediatric spinal cord injury. J Pediatr Rehabil Med. 2013;6(1):45-52. doi: 10.3233/PRM-130236. PMID 23481891
- [Result] Hwang M, Zebracki K, Betz RR, Mulcahey MJ, Vogel LC. Normative blood pressure and heart rate in pediatric spinal cord injury. Top Spinal Cord Inj Rehabil. 2013 Spring;19(2):87-95. doi: 10.1310/sci1902-87. PMID 23671378